CLINICAL TRIAL: NCT06920771
Title: A Randomized, Double-Blind, Placebo-Controlled, Multi-Centre Study to Assess the Efficacy of PURETHAL Mites Mixture 50,000 AUeq/mL Subcutaneous Immunotherapy in Adult Subjects With Moderate to Severe Allergic Rhinitis/Rhinoconjunctivitis With or Without Asthma Induced by House Dust Mite
Brief Title: A Randomized, Double-Blind, Placebo-Controlled, Multi-Centre Study to Assess the Efficacy of PURETHAL Mites Mixture 50,000 AUeq/mL Subcutaneous Immunotherapy in Adult Subjects With Moderate to Severe Allergic Rhinitis/Rhinoconjunctivitis With or Without Asthma Induced by House Dust Mite (HDM)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: HAL Allergy (Industry)
Collaborators: Ergomed (Industry); ClinCompetence Cologne GmbH (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PM/0059; 2023-504942-75-01 (EU CTIS Number)
Record Dates: First submitted 2024-10-18; First posted 2025-04-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2024-10

CONDITIONS: House Dust Mite Allergy; House Dust Mite Rhinitis
Keywords: PM0059; House dust mite; House dust mite allergy; House dust mite rhinitis; allergy; rhinitis; total nasal symptom score; TNSS; subcutaneous; Purethal
MeSH Terms: conditions — Dust Mite Allergy; Hypersensitivity; Rhinitis | interventions — Biological Products

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo Comparator: placebo (Placebo Comparator): Increasing volumes of placebo, will be administered by subcutaneous injection (starting with 0.05 ml) at weekly intervals till the maintenance dose (0.5 ml) is reached. Subsequently, maintenance dosages, corresponding to 0.5 ml of placebo, are given at 4-weekly intervals.
  Interventions: Biological: PURETHAL Mites 50,000 AUeq/ml; Biological: Biological/Vaccine: Placebo
- Experimental: PURETHAL Mites, 50,000 AU/ml (Active Comparator): Increasing dosages, corresponding to increasing volumes of drug solution (starting with 0.05 ml), will be administered by subcutaneous injection at weekly intervals till the maintenance dose (0.5 ml) is reached. Subsequently, maintenance dosages, corresponding to 0.5 ml of drug solution, are given at 4-weekly intervals.
  Interventions: Biological: PURETHAL Mites 50,000 AUeq/ml; Biological: Biological/Vaccine: Placebo

INTERVENTIONS:
Biological: PURETHAL Mites 50,000 AUeq/ml — Biological/Vaccine: Placebo
  Increasing volumes of placebo, will be administered by subcutaneous injection (starting with 0.05 ml) at weekly intervals till the maintenance dose (0.5 ml) is reached. Subsequently, maintenance dosages, corresponding to 0.5 ml of placebo, are given at 4-weekly intervals
Biological: Biological/Vaccine: Placebo — Increasing dosages, corresponding to increasing volumes of drug solution (starting with 0.05 ml), will be administered by subcutaneous injection at weekly intervals till the maintenance dose (0.5 ml) is reached. Subsequently, maintenance dosages, corresponding to 0.5 ml of drug solution, are given at 4-weekly intervals.

SUMMARY:
Rationale: Allergic rhinitis/rhinoconjunctivitis (ARC) is a global health problem, affecting 10-25% of the population. Allergen-specific immunotherapy is the only disease-modifying therapeutic option for subjects with house dust mites (HDM)-induced allergic rhinitis/rhinoconjunctivitis. This Phase 3 clinical study aims to demonstrate the effecacy of PURETHAL Mites (PM) Mixture subcutaneous immunotherapy (SCIT) compared to a placebo over one year of treatment in patients with moderate to severe HDM- induced allergic rhinitis/rhinoconjunctivitis (ARC), while also prioritizing the safety of the treatment. PM Mixture is a suspension of chemically modified extract from the house dust mites Dermatophagoides pteronyssinus (D. pter) and Dermatophagoides farinae (D. far), adsorbed to aluminium hydroxide. Modified extracts (allergoids) are associated with reduced allergenicity but with preserved immunogenicity. Based on the previous studies the dose of 0.5 mL of PM Mixture solution with concentration 50,000 AUeq/mL (allergen units in millilitre) was selected for this Phase 3 clinical study.

Objectives: The primary objective is to assess the efficacy of PM Mixture 50,000 AUeq/mL (0.5 mL) SCIT based on an average Total Combined Rhinitis Score (TCRS), which will be compared between PM Mixture and placebo groups. The TCRS consists of rhinitis symptom score and medication score measured daily over the last 8 weeks of the 1 year treatment.

Other secondary efficacy parameters will be compared between treatment groups to show efficacy: rhinitis symptom and medication scores separately as well as a combined symptom and medication score for nasal symptoms only (CSMS(n)); Total Combined Conductivities Score; nasal provocation test; immunological blood markers such as immunoglobulins E, G and G4; and Rhinitis Quality of Life Questionnaire (standardised) (RQLQ(S)).

Trial design: This is a randomized, double-blind, placebo controlled multi-centre clinical trial where subjects are participating for about 14 months.

Trial population: Patients (18-65 years of age) suffering from moderate to severe ARC induced by HDM with or without controlled asthma can be included in the study. The main criteria to evaluate the HDM allergy will be done by the following parameters: allergic medical history to HDM minimum 1 year; positive skin prick test and nasal provocation test HDM D. pter and/or D. far; certain level of allergen-specific immunoglobulin E to D. pter or D. far, and most importantly they should have sufficient rhinitis symptom score measured during 2 weeks at screening. Additionally patients should have sufficient lung functions confirmed by the spirometry, they may have asthma which should be controlled. Patients with a chronic or acute disease that might place the subject at an additional risk will not be included. Certain medications which can interfere with the study treatment or increase the health risks should be washed-out and can not be taken during the study.

Approximately 920 HDM-allergic subjects will be screened in order after the screening period to enroll 552 subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Prior to screening, subjects need to have signed the current approved Informed Consent Form (ICF).
2. Male or female subjects age 18-65 years at the time of informed consent.
3. Clinical history consistent with moderate-severe HDM allergic rhinitis (with or without asthma) according to the ARIA classification (Allergic Rhinitis and its Impact on Asthma) (Bousquet et al., 2008), for at least one year prior to the first dosing.
4. Subjects should be able and willing to complete daily e-Diaries for a period of 4 weeks during the screening period, 1 week after maintenance visit 7, and for a period of 8 weeks at the end of treatment under the same living conditions.
5. Forced Expiratory Volume 1 (FEV1) > 70% at Screening.
6. If a subject is asthmatic, asthma must be clinically controlled for at least three months before the screening using inhaled steroids and / or Long Acting Beta Agonists (corresponding to GINA treatment steps 1 -3) and inhaled steroid use should be on a stable, not higher dose than of ≤400 µg budesonide per day or dose-equivalent (≤500 µg beclometasone dipropionate; ≤160 µg ciclesonide;

   ≤250 µg fluticasone propionate; ≤200 µg mometasone furoate). Patients with asthma should use their standard asthma medication throughout the whole study period to ensure their asthma remains controlled.
7. Positive SPT to D. pter and/or D. far (mean wheal diameter ≥ 3 mm, negative control should be < 2 mm, histamine positive control should be ≥ 3 mm), assessed at Screening.
8. Subjects with a positive NPT for D. pter extract at Screening (Lebel score ≥6 at 10,000 AU/mL, test should be postponed, if baseline score is ≥ 3 or if negative control score is > 3).
9. Allergen specific serum IgE level for D. pter and/or D. far of > 0.7 U/mL, assessed at Screening.
10. Subjects need to have an average daily TNSS of at least 8 out of 12 points at baseline, determined according to the daily e-Diary entries during 2 weeks of baseline assessment. Subjects should have a minimum e-Diary entry compliance of 70% for which the average is calculated.
11. Negative serum pregnancy test at screening for women of childbearing potential.
12. Females of childbearing potential must be using highly effective and acceptable methods of birth control (as per the CTFG recommendations) to prevent pregnancy and agree to continue to practice an acceptable method of contraception for the duration of participation in the trial. Contraceptive measures considered adequate are:

    1. combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal)
    2. progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable)
    3. intrauterine device (IUD)
    4. intrauterine hormone-releasing system (IUS)
    5. bilateral tubal occlusion
    6. vasectomised partner
    7. sexual abstinence Waivers to the inclusion criteria will NOT be allowed.

Exclusion Criteria:

1. A clinically relevant history of symptomatic seasonal ARC and/or a positive SPT (mean wheal diameter ≥ 3 mm) caused by an allergen (including animal hair and dander), to which the subject is regularly exposed and/or exposure is overlapping with the e-Diary completion periods at Screening and at the end of treatment.
2. Nasal surgery and/or severe nasal or severe oral disease within 6 months prior to Screening.
3. Patients not adhering to the e-Diary procedure and/or procedure for Rescue Medication use during e-Diary phase.
4. Severe asthma (GINA 2022 treatment steps 4 - 5).
5. Uncontrolled asthma, as defined by any of the following:

   1. Asthma Control Test (ACT) ≤19,
   2. FEV1 ≤70% of predicted value,
   3. Emergency room visit for asthma attack/exacerbation within 6 months prior to screening,
   4. At least 1 hospitalization due to asthma within the last year,
   5. History of intubation/mechanical ventilation due to asthma,
   6. More than 2 courses of oral steroids used for treatment of asthma within the last 6 months prior to Screening,
   7. Daily use of inhaled corticosteroids >400mcg budesonide or equivalent.
6. History of anaphylaxis with cardio-respiratory symptoms (food allergy, drugs or an idiopathic reaction).
7. Previous treatment with AIT with HDM allergen or a cross-reacting allergen for more than 1 month at the maintenance level within the last 5 years. Initiation of HDM SCIT is acceptable, if treatment has been discontinued before reaching maintenance dose.
8. AIT (subcutaneous, sublingual or oral) with other allergens than HDM within the last 3 months prior to screening or planned during the trial period.
9. Participation in a clinical trial within the last 3 months prior to screening (e.g.

new investigational drug or biological) or during the trial. 10. Any vaccination (including COVID-19) less than 1 week prior to screening, during screening and the up-dosing phase and the TCRS scoring periods. 11. Any immunosuppressive treatment or anti-IgE therapy within the last 6 months prior to the first dosing of the trial drug and during the trial 12. Any treatment with β-adrenergic blockers unless prescribed as per treatment standards to the subject if the medical benefit will prevail the risks upon investigators discretion. 13. Hypersensitivity to any of the other components of the investigational product. 14. Severe immune disorders (including autoimmune diseases) and/or diseases requiring immunosuppressive medication. 15. Active COVID-19 infection at the time of screening or 2 weeks before. 16. Active malignancies or any malignant disease in the last 5 years. 17. A chronic or acute disease that in the opinion of the investigator might place the subject at an additional risk, including but not limited to the following: cardiovascular insufficiency, any severe or unstable lung diseases, endocrine disorders, clinically significant renal or hepatic diseases, haematological disorders, severe atopic dermatitis, other relevant skin diseases (affecting SPT testing areas). 18. Diseases with a contraindication for the use of adrenaline/epinephrine (e.g.

hyperthyroidism, glaucoma). 19. Use of prohibited medication and/or not able to discontinue medications that are prohibited during the specified trial periods. 20. Moderate to severe nasal obstructive disease such as polyps, septum deviation. 21. Clinically significant chronic sinusitis or ocular infection. 22. Female subjects of childbearing potential who are pregnant or lactating. 23. Alcohol, drug, or medication abuse within the past year and during the trial.

24. Any (expected) lack of cooperation or compliance upon the discretion of the investigator. 25. Severe psychiatric, psychological, or neurological disorders. 26. Employees of the Sponsor, CRO, clinical study site and/or who are 1st grade relatives, or partners of the investigator. 27. Known commitment to an institution by virtue of an order issued either by the judicial or the administrative authorities 28. Expected changes in average HDM exposure during the trial (e.g. new avoidance measures, relocation and holidays or trips lasting more than 10 days during the efficacy assessment period)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 552 (Estimated)
Dates: Start 2024-09-09 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Primary objective | Last 8 weeks (before end of study) of the intervention.
  To assess clinical efficacy of PM Mixture 50,000 AUeq/mL (0.5 mL) SCIT in subjects suffering from moderate to severe HDM-induced ARC, measured by difference in the average Total Combined Rhinitis Score (TCRS) during the last 8 weeks of one (± 1 month) year treatment, between PM treatment and placebo.
  Each symptom will be individually graded and then summed to a maximum of 24 points.

SECONDARY OUTCOMES:
To assess the effect of PM treatment by comparing the average daily Total Nasal Symptom Score (TNSS) between PM and placebo during the last 8 weeks of one (± 1 month) year treatment of subjects with HDM-allergic ARC. | The last 8 weeks of one (± 1 month) year treatment.
  To assess the effect of PM treatment by comparing the average daily Total Nasal Symptom Score (TNSS) between PM and placebo during the last 8 weeks of one (± 1 month) year treatment of subjects with HDM-allergic ARC.

CONTACTS AND LOCATIONS:
Overall Officials: Hans Hoogeveen, Study Director — Head of Clinical Development
Locations (68):
- Bulgaria (6):
  - UMBAL Kaspela, Plovdiv
  - Medical Center Prolet EOOD, Rousse
  - Medical Center Smolyan, Smolyan
  - DCC Convex, Sofia
  - Diagnostic-Consulativ Senter Ascendent, Sofia
  - University Hospital Alexandrovska, Sofia
- Germany (19):
  - Emovis GmbH, Berlin
  - Praxis Dr. Ginko, Bonn
  - Praxis Dr. Elke Decot, Dreieich
  - HNO-Praxis Dr. Udo Schäfer, Dresden
  - HNO Praxis Dr. Uta Thieme, Duisburg
  - Medizentrum Essen-Borbeck, Essen
  - Pneumologisches Forschungsinstitut Hohegeest GbR, Geesthacht
  - HNO-Facharztpraxis Alte Post, Göttingen
  - HNO Research GmbH, Itzehoe
  - Hospital Schleswig-Holstein. Klinik für Dermatologie, Venerologie und Allergologie., Kiel
  - BAG Prof. G. Hoheisel/Dr. A. Bonitz Praxis für Pneumologie und Allergologie - Studienzentrum, Leipzig
  - Praxis Dr. Bohn, Mittweida
  - Ballenberger, Freytag, Wenisch -Institut für klinische Forschung GmbH, Neu-Isenburg
  - Studienzentrum MOL BAG Dres. E.Hippke & S. Runge, Neuenhagen
  - KliFOs - Klinische Forschung Osnabrück, Osnabrück
  - Studienzentrum Dr.Schlenska, Peine
  - Studienzentrum Dr.Laßmann, Saalfeld
  - Allergo GmbH - Prüfzentrum Schorndorf, Schorndorf
  - Klinikum Stuttgart - Krankenhaus Bad Cannstatt, Stuttgart
- Latvia (2):
  - LOR Clinic, Riga
  - The Center of Investigation in Treatment of Allergyc Diseases, Riga
- Lithuania (7):
  - CD8 clinic, Kaunas
  - Lithuanian University of Health Sciences Kauno klinikos, Kaunas
  - Inovatyvios alergologijos centras, Vilnius
  - JSC Center for Diagnosis and Treatment of Allergic Diseases, Vilnius
  - JSC Family Doctor, Vilnius
  - JSC Inlita, Vilnius
  - JSC Verkiu clinic, Vilnius
- Poland (34):
  - NZOZ Homeo Medicus Poradnia Alergologiczna, Bialystok
  - Prywatna Praktyka Lekarska Gabinet Pediatryczno-Alergologiczny Anna Płoszczuk, Bialystok
  - Specjalistyczna Praktyka Lekarska AlerMedica, Bialystok
  - Centrum Medyczne KERmed, Bydgoszcz
  - Pratia - Ośrodek Badań Klinicznych, Częstochowa
  - Clinica Vitae Spółka z o. o., Gdansk
  - Indywidualna Specjalistyczna Praktyka Lekarska Elżbieta Matusz, Gryfice
  - Centrum Medyczne Angelius Provita, Katowice
  - Specjalistyczna Praktyka Lekarska dr n.med. Joanna Orlicz-Widawska, Katowice
  - PZU Zdrowie Centra Medyczne Kielce, Kielce
  - Indywidualna Specjalistyczna Praktyka Lekarska Jan Zdanowski Specjalista Alergolog, Koszalin
  - Centrum Nowoczesnych Terapii "Dobry Lekarz" Sp. z o.o., Krakow
  - Krakowskie Centrum Medyczne Sp. z o.o - FutureMeds Kraków, Krakow
  - Małopolskie Centrum Alergologii sp z o.o., Krakow
  - Clinmedica Research sp. z o.o., Lodz
  - CM Szpital Św. Rodziny, Lodz
  - IP Clinic Sp. z o. o., Lodz
  - Medical University of Lodz, Lodz
  - Centrum Diagnostyczno-Terapeutyczne Medicus Sp. z o.o., Lubin
  - ALERGOTEST s.c. Specjalistyczne Centrum Medyczne, Lublin
  - Centrum Alergoologii Specjalistyczna Przychodnia Alergologiczna, Lublin
  - Pro Life Medica Sp. z o.o., Lublin
  - Uniwersytecki Szpital Kliniczny Nr 4 w Lublinie, Lublin
  - Centrum Alergologii, Poznan
  - NZOZ Alergo-Med, Poznan
  - Poradnie Specjalistyczne Alergologia Plus - Justyna Rakowicz, Poznan
  - NSZOZ Puls Med, Skarżysko-Kamienna
  - Alergo-Med Specjalistyczna Przychodnia Lekarska Sp. z o. o., Tarnów
  - Gabinet Lekarski Bożena Kubicka-Kozik, Tomaszów Mazowiecki
  - Centrum Alergologii Irmed Irena Wojciechowska, Warsaw
  - ETG Warszawa, Warsaw
  - POLIMEDICA CENTRUM BADAŃ, PROFILAKTYKI I LECZENIA Sp. z o.o. - POLIMEDICA PTG, Warsaw
  - All-Med - Specjalistyczna Opieka Medyczna - Medyczny Instytut Badawczy, Wroclaw
  - NZOZ Centrum Usług Medycznych "PROXIMUM" Sp. z o. o., Wroclaw

IPD SHARING:
Plan to Share IPD: No